CLINICAL TRIAL: NCT04550468
Title: Impact of a Low-carbohydrate Versus Low-fat Breakfast on Blood Glucose Control in Type 2 Diabetes
Brief Title: Low-carbohydrate Versus Low-fat Breakfast in Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: University of Wollongong (Other)
Responsible Party: Principal Investigator, Jonathan Little, Associate Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: H19-03179
Record Dates: First submitted 2020-07-15; First posted 2020-09-16 (Actual); Results first posted 2025-02-04 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-02

CONDITIONS: Dietary Habits
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-Carb High-Fat Breakfast (Experimental): Participants will follow a daily low carbohydrate high fat breakfast intervention for 3 months.
  Interventions: Other: Low-Carb High-Fat breakfast
- Low fat "Standard Care" Control Breakfast (Active Comparator): Participants will follow a daily low fat "standard care" control breakfast intervention for 3 months.
  Interventions: Other: Low fat "standard care" control breakfast

INTERVENTIONS:
Other: Low-Carb High-Fat breakfast — Participants will receive 8 low-carb high-fat breakfast meal recipes to follow daily during 3 months.
  Arms: Low-Carb High-Fat Breakfast
Other: Low fat "standard care" control breakfast — Participants will receive 8 low-fat breakfast meal recipes to follow daily during 3 months.
  Arms: Low fat "Standard Care" Control Breakfast

SUMMARY:
The prevalence of type 2 diabetes (T2D) is increasing worldwide, with ~380 M currently suffering from this chronic, debilitating disease. T2D is characterized by high blood glucose levels in the mornings and after meals. The largest hyperglycemic spike often occurs after breakfast. Targeting this meal may be a simple, feasible strategy to improve glycemic control and reduce risk for diabetes complications. It is hypothesized that consuming a low carbohydrate high fat (LCHF) breakfast for 3 months, when compared to a standard low-fat breakfast will improve blood glucose control, increase satiety and improve body composition in people with T2D. This information will test whether the simple dietary strategy of limiting carbohydrates at breakfast could help in managing T2D.

DETAILED DESCRIPTION:
A 3-month parallel-group randomized controlled trial will be conducted. Eligible participants will be randomized to either the Low-carb High-fat breakfast (LCHF, n=41) or a low-fat "standard care" control breakfast (CTL, n=41), to be consumed daily for a period of 3 months.

Due to COVID-19 pandemic, this study was adapted to be conducted remotely through video/telephone conference meetings between participants and study staff, along with mailing of study materials before and after the intervention for remote data collection.

Each group will be provided with a menu of 8 LCHF breakfasts or 8 CTL breakfasts from which to choose each morning. Breakfast options (designed by a registered dietitian) will be controlled in macronutrient content and calories (~400-500 kcal), but allow for personal preference and autonomy to promote adherence.

ELIGIBILITY:
Inclusion Criteria:

* physician-diagnosed T2D of ≥1 year;
* current HbA1c of < 8.5%;
* BMI: >25 kg/m2; (as of July 5, 2021, BMI cut off was expanded from 25-40 kg/m2 to higher than 25kg/m2 to facilitate recruitment)
* blood pressure of <160/99 mm Hg assessed according to guidelines;
* non-smoking;
* not on hormone replacement therapy, corticosteroids, or anti-inflammatory medications;
* 20-79 years old.

Exclusion Criteria:

* Use of exogenous insulin;
* taking more than 2 glucose lowering medications;
* ongoing medical treatment for diseases such as cancer, auto-immune or inflammatory disease, liver or kidney disorders;
* allergy, intolerance or aversion to eggs or any other dietary restrictions (e.g., vegan, breakfast skipping) that will prevent them from following the standardized study diets;
* being unable to follow remote guidance by internet or smartphone
* being unable to follow the controlled diet instructions;.

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of British Columbia, Kelowna, British Columbia, Canada

REFERENCES:
- [Derived] Oliveira BF, Chang CR, Oetsch K, Falkenhain K, Crampton K, Stork M, Hoonjan M, Elliott T, Francois ME, Little JP. Impact of a Low-Carbohydrate Compared with Low-Fat Breakfast on Blood Glucose Control in Type 2 Diabetes: A Randomized Trial. Am J Clin Nutr. 2023 Jul;118(1):209-217. doi: 10.1016/j.ajcnut.2023.04.032. Epub 2023 May 29. PMID 37257563

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 121 were included in analysis according to intention-to-treat principle
Groups:
- Low-Carb High-Fat Breakfast: Participants followed a daily low carbohydrate high fat breakfast intervention for 3 months.
  Low-Carb High-Fat breakfast: Participants received 8-10 low-carb high-fat breakfast meal recipes to follow daily during 3 months.
- Low Fat "Standard Care" Control Breakfast: Participants followed a daily low fat "standard care" control breakfast intervention for 3 months.
  Low fat "standard care" control breakfast: Participants received 8 low-fat breakfast meal recipes to follow daily during 3 months.
Period: Overall Study
Arm/Group | Low-Carb High-Fat Breakfast | Low Fat "Standard Care" Control Breakfast
Started | 64 | 63
Completed | 45 | 48
Not Completed | 19 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low-Carb High-Fat Breakfast | Low Fat "Standard Care" Control Breakfast | Total
Number analyzed (Participants) | 60 | 61 | 121
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (9) | 64 (10) | 64 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 35 | 64
  Male | 31 | 26 | 57
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 38 | 37 | 75
  Australia | 22 | 24 | 46
Duration of T2D, mean (SD), years [Mean (Standard Deviation); unit: years] | 10 (8) | 9 (6) | 9 (7)
HbA1c (%) [Mean (Standard Deviation); unit: percent] | 6.9 (0.8) | 7.0 (0.7) | 7.0 (0.7)
Weight (kg) [Mean (Standard Deviation); unit: kilograms] | 95.8 (26.3) | 90.8 (18.8) | 93.3 (22.9)
BMI (kg/m2) [Mean (Standard Deviation); unit: kg/m2] | 33.2 (8.2) | 31.4 (6.2) | 32.3 (7.3)
Waist Circumference (cm) [Mean (Standard Deviation); unit: centimeters] | 111.1 (16.2) | 109.6 (15.7) | 110.2 (15.9)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Hemoglobin A1c at 12 Weeks
Description: Hemoglobin A1c measured at baseline and after 12 weeks of following the low-carbohydrate breakfast or low-fat breakfast
Time Frame: Baseline to 12 weeks of diet
Measure: Mean (95% Confidence Interval); unit: % of HbA1c
Arm/Group | Low-Carb High-Fat Breakfast | Low Fat "Standard Care" Control Breakfast
Number analyzed (Participants) | 60 | 61
% of HbA1c | -0.3 [-0.4 to -0.1] | -0.1 [-0.2 to 0.1]

2. Secondary Outcome: Change From Baseline Fasting Blood Glucose at 12 Weeks
Description: Mean fasting blood glucose from 14 days measured at baseline and after 12 weeks of following the low-carbohydrate breakfast or low-fat breakfast
Time Frame: Mean values for the first 14 days (weeks 1-2) and mean values for the last 14 days (weeks 11-12) of the intervention
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Low-Carb High-Fat Breakfast | Low Fat "Standard Care" Control Breakfast
Number analyzed (Participants) | 60 | 61
mmol/L
  First 14 days | 7.0 (1.3) | 7.6 (1.9)
  Last 14 days | 7.0 (1.3) | 7.6 (1.7)

3. Secondary Outcome: Change From Baseline Fasting Blood Insulin at 12 Weeks
Description: Average fasting blood insulin measured at baseline and after 12 weeks of following the low-carbohydrate breakfast or low-fat breakfast
Time Frame: Baseline to 12 weeks of diet
Population: Due to logistics and budget, samples were not collected for insulin measurement.
Arm/Group | Low-Carb High-Fat Breakfast | Low Fat "Standard Care" Control Breakfast
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change From Baseline Blood Lipids at 12 Weeks
Description: Mean triglycerides, total, HDL, and LDL cholesterol at baseline and after 12 weeks of following the low-carbohydrate breakfast or low-fat breakfas
Time Frame: Baseline to 12 weeks of diet
Population: Blood samples were not collected for triglycerides.
Measure: Mean (95% Confidence Interval); unit: % change
Arm/Group | Low-Carb High-Fat Breakfast | Low Fat "Standard Care" Control Breakfast
Number analyzed (Participants) | 60 | 61
% change
  Total cholesterol | -0.3 [-9.1 to 8.5] | -5.9 [-13.8 to 2.0]
  HDL cholesterol | -3.6 [-7.3 to 0.1] | -3.8 [-7.4 to -0.2]
  cholesterol/HDL ratio | 13 [0 to 28] | 6 [-6 to 19]
  non-HDl cholesterol | 5.9 [-2.7 to 14.5] | -1.9 [-9.8 to 6]
  Triglycerides: number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change From Baseline Inflammation Marker High Sensitive Reactive Protein (hsCRP) at 12 Weeks
Description: Blood inflammation marker (hsCRP) at baseline and after 12 weeks of following the low-carbohydrate breakfast or low-fat breakfast
Time Frame: Baseline to 12 weeks of diet
Measure: Mean (95% Confidence Interval); unit: % change
Arm/Group | Low-Carb High-Fat Breakfast | Low Fat "Standard Care" Control Breakfast
Number analyzed (Participants) | 60 | 61
% change | 10 [-15 to 42] | -6 [-27 to 21]

6. Secondary Outcome: Hunger/Satiety Levels
Description: Levels of hunger and satiety measured by a 0 to 100 millimeter visual analog scale [ranges across a continuum from none (0) to an extreme amount (100) of Hunger, Satiety, Fullness, Appetite] How hungry do you feel? How satisfied do you feel? How full do you feel? How much food do you think you can eat?
Time Frame: Weeks 1, 6 and 12
Measure: Mean (Standard Deviation); unit: score on a scale (mm)
Arm/Group | Low-Carb High-Fat Breakfast | Low Fat "Standard Care" Control Breakfast
Number analyzed (Participants) | 60 | 61
score on a scale (mm)
  How hungry do you feel? week 1 | 22 (18) | 27 (23)
  How satisfied do you feel? week 1 | 69 (17) | 70 (19)
  How full do you feel? week 1 | 72 (21) | 69 (23)
  How much food do you think you can eat? week 1 | 46 (25) | 47 (25)
  How hungry do you feel? week 6 | 26 (21) | 26 (22)
  How satisfied do you feel? week 6 | 65 (21) | 65 (22)
  How full do you feel? week 6 | 72 (19) | 67 (22)
  How much food do you think you can eat? week 6 | 49 (24) | 46 (25)
  How hungry do you feel? week 12 | 29 (25) | 26 (23)
  How satisfied do you feel? week 12 | 64 (21) | 64 (22)
  How full do you feel? week 12 | 70 (22) | 66 (23)
  How much food do you think you can eat? week 12 | 48 (23) | 43 (25)

7. Secondary Outcome: Dietary Intake
Description: Dietary calorie intake assessed by three 3-day food records during the 12-week intervention
Time Frame: Mean dietary intake assessed during the 12-week intervention
Measure: Mean (Standard Deviation); unit: kilocalories
Arm/Group | Low-Carb High-Fat Breakfast | Low Fat "Standard Care" Control Breakfast
Number analyzed (Participants) | 60 | 61
kilocalories
  total energy | 1701 (510) | 1927 (480)
  total carbohydrate energy | 601 (225) | 883 (288)
  total protein energy | 347 (102) | 325 (112)
  total fat energy | 753 (251) | 719 (255)

8. Secondary Outcome: Change From Baseline Body Weight at 12 Weeks
Description: Body weight measured in kilograms at baseline and after 12 weeks of following the low-carbohydrate breakfast or low-fat breakfast
Time Frame: Baseline to 12 weeks of diet
Measure: Mean (95% Confidence Interval); unit: % change
Arm/Group | Low-Carb High-Fat Breakfast | Low Fat "Standard Care" Control Breakfast
Number analyzed (Participants) | 60 | 61
% change | -1.2 [-2.3 to -0.1] | -0.9 [-1.9 to 0.1]

9. Secondary Outcome: Change From Baseline Body Mass Index at 12 Weeks
Description: Body mass Index measured in weight in kilograms divided by the square of height in meters at baseline and after 12 weeks of following the low-carbohydrate breakfast or low-fat breakfast
Time Frame: Baseline to 12 weeks of diet
Measure: Mean (95% Confidence Interval); unit: %change
Arm/Group | Low-Carb High-Fat Breakfast | Low Fat "Standard Care" Control Breakfast
Number analyzed (Participants) | 60 | 61
%change | -1.2 [-2.3 to -0.1] | -1.1 [-2.2 to 0.0]

10. Secondary Outcome: Continuous Glucose Monitoring
Description: Measures of overall glucose control by continuous glucose monitoring device
Time Frame: Mean values for the first 14 days (weeks 1-2) and mean values for the last 14 days (weeks 11-12) of treatment
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Low-Carb High-Fat Breakfast | Low Fat "Standard Care" Control Breakfast
Number analyzed (Participants) | 60 | 61
mmol/L
  Fasting glucose first 14 days | 6.5 (1.5) | 6.5 (1.5)
  Fasting glucose last 14 days | 7.0 (1.9) | 6.8 (1.7)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Low-Carb High-Fat Breakfast | Low Fat "Standard Care" Control Breakfast
All-Cause Mortality (participants affected / at risk) | 0/64 | 0/63
Serious Adverse Events (participants affected / at risk) | 0/64 | 0/63
Other Adverse Events (participants affected / at risk) | 0/64 | 0/63

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-10-01): https://cdn.clinicaltrials.gov/large-docs/68/NCT04550468/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-23): https://cdn.clinicaltrials.gov/large-docs/68/NCT04550468/SAP_001.pdf